CLINICAL TRIAL: NCT03759652
Title: Surveillance of Surgical Site Infections and Non-surgical Infections of Neurosurgical Patient. Retrospective Before-after Cohort Study at a Tertiary Care Hospital in Poland
Brief Title: Surgical and Non-surgical Infections of Neurosurgical Patient: Before-after Cohort Study
Status: Completed | Type: Observational
Sponsor: Polskie Towarzystwo Zakażeń Szpitalnych (Other)
Responsible Party: Sponsor
Other Study IDs: PTZS Neurosurgery 2018
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Neurosurgery
Keywords: neurosurgery; surgical site infections; spinal surgery; craniotomy; laminectomy
MeSH Terms: conditions — Surgical Wound Infection | interventions — Controlled Before-After Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infected, before-after studyt: 2003: neurosurgical patients; 2003: the beggining of active and target HAI surveillance
  Interventions: Behavioral: before-after study
- infected, before-after studyt: 2017: neurosurgical patients; 2017: the effective of active and target HAI surveillance
  Interventions: Behavioral: before-after study

INTERVENTIONS:
Behavioral: before-after study — The data analysed involve the time when the targeted, active surveillance of infections was establised, initially: 2003-2017, using tools (definitions, protocols) in accordance with the National Healthcare Safety Network (NHSN), then from 2012, HAI recognition methodology and HAI record-keeping has followed the Surveillance Network (HAI-Net), European Centre for Disease Prevention and Control (ECDC).

SUMMARY:
Continuous surveillance in 2003-2017 allowed to detect HAIs in patients staying in a 42-bed neurosurgery unit with 6 intensive neurosurgical supervision beds. 10,332 surgical patients were qualified for the study. The study was carried out in the framework of a national surveillance of HAI programme following methodology recommended by Healthcare-Associated Infections Surveillance Network (HAI-Net), European Centre for Disease Prevention and Control. Intervention in this before-after study (2003-2017) comprised standardised surveillance of HAI with regular analysis and feedback.

DETAILED DESCRIPTION:
Supervision of HAIs was carried out in the neurosurgery unit in 2003-2017 in St. Luke Provincial Hospital in Tarnów, Poland. The department offers 42 hospital beds (including 6 intensive supervision beds, where mechanical ventilation is also used). Patients in very poor clinical condition do not stay in this department as they are generally sent to a separate general intensive care unit. Active surveillance of infections was implemented in the hospital in 2001 and the experiences concerning the neurosurgery unit were already the subject of previous general analyses not including trend analysis or detailed analyses of various HAI clinical forms [Wałaszek NCH 2015]. The Infection Control Team consists of a doctor, who is employed on a 1/3 full-time equivalent basis and 4 full-time epidemiological nurses.

The data analysed involve the time when the unit in question began targeted, active surveillance of infections, initially: 2003-2012, using tools (definitions, protocols) in accordance with the National Healthcare Safety Network (NHSN) [Emori, NNIS], then from 2012, HAI recognition methodology and HAI record-keeping has followed the Surveillance Network (HAI-Net), European Centre for Disease Prevention and Control (ECDC) [ECDC 4.3, 2012; HAI-Net ICU 1.02. ECDC; 2015]. For the purposes of this analysis, HAI cases originally qualified in 2002-2012 according to the NHSN criteria were retrospectively subjected to reclassification according to the ECDC definitions from 2012 (they concerned BSI, PN and UTI), hence, all HAI cases were qualified into individual HAI categories according to the ECDC case definition keeping the division into: catheter-related BSI and BSI secondary to another infection, five subcategories of PN and three forms of SSI. The surgeries performed were stratified by type of operation conforming to the International Classification of Procedures in Medicine ICD 9-CM, according to the NHSN code (International Classification of Diseases) (Supplementarty Material, Table 1).

Beginning in 2003, changes were being implemented as regards supervision of infections by the Infection Control Team together with the staff of the departments (neurosurgery, operating block and infection control team), which encompassed, among others:

1. hospital admission rules for shortening of the pre-operative stay and optimal patient preparation for surgery to limit emergency surgery; preparation of the surgical team
2. work organization of the operating block: among others, preoperative checklist, surgical hand hygiene, preparation of the operating field and surgical drape, application of antiseptic to the edges of the wound before sewing it;
3. perioperative procedure: patient preparation for surgery, among others, bathing the patient immediately prior to surgery, hair removal, changing the bed linen and patient's clothing immediately before surgery, patient care during the postoperative period, and above all, the 5 moments for hand hygiene and post-operative dressing and wound control.

In addition: regular analysis and feedback have also been implemented.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of neurosurgical disorders
* requiring surgery

Exclusion Criteria:

patients without surgery intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery in the Neurosurgery Ward in St. Luke Provincial Hospital in Tarnów, Poland, in 2003-2017
Sampling Method: Non-Probability Sample
Enrollment: 10332 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
incidence of surgical site infection | 2003-2017
  the cumulative incidence of surgical site infection (SSI) was calculated by dividing the number of SSI cases by the number of patients undergoing surgery and multiplying by 100
incidence of pneumonia | 2003-2017
  the cumulative incidence of post-procedure pneumonia was calculated by dividing the number of pneumonia cases by the number of patients undergoing surgery and multiplying by 100
incidence of bloodstream infections | 2003-2017
  the cumulative incidence of bloodstream infections (BSI) was calculated by dividing the number of BSI cases by the number of patients undergoing surgery and multiplying by 100

CONTACTS AND LOCATIONS:
Overall Officials: Jadwiga Wójkowska-Mach, Principal Investigator — Jagiellonian University Medical School
Locations (1):
- Jagiellonian University Medical School, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No